CLINICAL TRIAL: NCT00084578
Title: A Randomized Trial of Celecoxib and Rosiglitazone, Alone and in Combination, in Patients With Early Stage Non-Invasive Bladder Carcinoma Undergoing Cystoscopic Surveillance and in Patients With Muscle-Invasive Bladder Cancer Undergoing Radical Cystectomy
Brief Title: Celecoxib and Rosiglitazone in Treating Patients Who Are Undergoing Cystoscopic Surveillance for Early-Stage Noninvasive Carcinoma of the Bladder or Radical Cystectomy for Muscle-Invasive Carcinoma of the Bladder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to drug toxicity
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: FCCC-03018; CDR0000365460 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; stage I bladder cancer; stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Celecoxib; Rosiglitazone; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: celecoxib
Drug: rosiglitazone maleate
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Celecoxib may stop the growth of tumor cells by blocking the enzymes necessary for their growth and by stopping blood flow to the tumor. Rosiglitazone may help tumor cells develop into normal bladder cells.

PURPOSE: This randomized clinical trial is studying how well giving celecoxib together with rosiglitazone works in treating patients who are undergoing cystoscopic surveillance (screening) for early-stage noninvasive (carcinoma in situ) carcinoma (cancer) of the bladder or radical cystectomy for muscle-invasive carcinoma (cancer has spread into the muscle layer of bladder tissue) of the bladder.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether rosiglitazone and celecoxib, administered alone or in combination, cause changes in the expression of effector molecules, peroxisome proliferator-activated receptor-γ (PPAR-γ) and cyclo-oxygenase-1 (COX-1), in patients with early-stage non-invasive carcinoma of the bladder undergoing cystoscopic surveillance or in patients with muscle-invasive carcinoma of the bladder undergoing radical cystectomy.

Secondary

* Determine whether these regimens result in changes in the expression of downstream effector molecules that mediate cellular proliferation and apoptosis in these patients.
* Determine the relationship between tissue levels of biomarkers of drug effect, proliferation, and apoptosis and the systemic biomarkers of response to treatment, in terms of COX-2 activity and the levels of the endogenous PPAR-γ ligand, in patients treated with these regimens.
* Determine the toxicity of these regimens in these patients.
* Determine the frequency of recurrence and the time to progression in patients undergoing cystoscopic surveillance.

OUTLINE: This is a randomized, pilot, cohort study. Patients are assigned to 1 of 2 cohorts according to disease stage (Ta, Tis, T1, N0, M0 vs T2-4, NX, M0).

* Stage 1:

  * Cohort 1: Patients receive oral celecoxib twice daily and oral rosiglitazone once daily for 1 year in the absence of disease progression or unacceptable toxicity.
  * Cohort 2: Patients receive oral celecoxib twice daily and oral rosiglitazone once daily for 14 days. Patients then undergo cystectomy.
* Stage 2: Patients are randomized into 1 of 2 treatment arms.

  * Arm I:

    * Cohort 1: Patients receive oral celecoxib twice daily for 1 year in the absence of disease progression or unacceptable toxicity.
    * Cohort 2: Patients receive oral celecoxib twice daily for 14 days. Patients then undergo cystectomy.
  * Arm II:

    * Cohort 1: Patients receive oral rosiglitazone once daily for 1 year in the absence of disease progression or unacceptable toxicity.
    * Cohort 2: Patients receive oral rosiglitazone once daily for 14 days. Patients then undergo cystectomy.

Patients in cohort 1 (in both stages) undergo cystoscopic surveillance every 3 months.

PROJECTED ACCRUAL: A total of 120 patients (20 per cohort in study stage 1; 40 per treatment arm [20 per cohort in each arm] in study stage 2) will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and clinically confirmed bladder cancer

  * Cohort 1

    * Papillary transitional cell carcinoma of the urinary bladder

      * Stage Ta or T1 (grade 1 or 2), N0, M0 disease
      * Must have undergone complete transurethral resection of the bladder within the past 28 days AND/OR
    * Carcinoma in situ of the urinary bladder

      * Stage Tis, N0, M0 disease
      * Must have undergone biopsy within the past 28 days
    * No histological and pathological evidence of invasion of the underlying muscle (stage T2)
  * Cohort 2

    * Muscle-invasive papillary transitional cell carcinoma of the urinary bladder
    * Stage T2-4, NX, M0 disease
    * Intending to undergo radical cystectomy
    * Must have had an upper tract (ureter and renal pelvic) evaluation by intravenous pyelogram, CT scan, or MRI that proved normal within the past year

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC > 4,000/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin < 2 times upper limit of normal (ULN)
* SGOT and SGPT < 3 times ULN

Renal

* Creatinine ≤ 2.5 mg/dL

Other

* No other malignancy within the past 3 years except non-invasive bladder cancer, adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix
* No history of uncontrolled peptic ulcer disease
* No history of unexplained hypoglycemia
* No known sensitivity to celecoxib or rosiglitazone
* No allergy to sulfonamides
* No history of asthma, urticaria, or allergic reaction after taking aspirin or other NSAIDs
* No underlying uncontrolled medical illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 months since prior intravesical BCG

Chemotherapy

* No prior intravesical or systemic chemotherapy

Endocrine therapy

* No concurrent insulin

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Other

* At least 2 weeks since prior use of non-steroidal anti-inflammatory drugs (NSAIDs) (including COX-2 inhibitors) for more than 3 consecutive days except low-dose (81 mg) aspirin
* No concurrent beta-blockers
* No concurrent NSAIDs
* No other concurrent oral hypoglycemic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lewis, MD, Principal Investigator — Fox Chase Cancer Center